CLINICAL TRIAL: NCT00526110
Title: A Phase I/II Study of Docetaxel, 5-Fluorouracil and Oxaliplatin (D-FOX) in Patients With Untreated Locally Unresectable or Metastatic Adenocarcinoma of the Stomach or Gastroesophageal Junction
Brief Title: Docetaxel, 5-Fluorouracil and Oxaliplatin in Adenocarcinoma of the Stomach or Gastroesophageal Junction Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Sanofi-Synthelabo (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2004-0290; NCI-2010-00750 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2007-09-04; First posted 2007-09-06 (Estimated); Results first posted 2016-10-31 (Estimated); Last update posted 2016-10-31 (Estimated); Status verified 2016-09

CONDITIONS: Gastrointestinal Diseases
Keywords: Gastrointestinal Diseases; Adenocarcinoma of the Stomach; Gastroesophageal Junction Cancer; Cancer of the Stomach; 5-Fluorouracil; 5-FU; Adrucil; Efudex; Docetaxel; Oxaliplatin; Eloxatin; Taxotere; Esophagus
MeSH Terms: conditions — Gastrointestinal Diseases; Stomach Neoplasms | interventions — Fluorouracil; Docetaxel; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 5-Fluorouracil + Docetaxel + Oxaliplatin (Experimental): 5-Fluorouracil 2.2 Gm/m^2 intravenously (IV) over 48 hours on Day 1. Docetaxel 20 mg/m^2 IV over 60 minutes. Oxaliplatin 85 mg/m^2 IV over 120 minutes on Day 1.
  Interventions: Drug: 5-Fluorouracil; Drug: Docetaxel; Drug: Oxaliplatin

INTERVENTIONS:
Drug: 5-Fluorouracil — 2.2 Gm/m^2 IV over 48 hours on Day 1.
  Other Names: 5-FU; Adrucil; Efudex
Drug: Docetaxel — 20 mg/m^2 IV over 60 minutes
  Other Names: Taxotere
Drug: Oxaliplatin — 85 mg/m^2 IV over 120 minutes on Day 1.
  Other Names: Eloxatin

SUMMARY:
Phase I Objectives

Primary:

1. The primary objective of this study is to determine the maximum tolerated dose (MTD) of Docetaxel combined with 5-Fluorouracil and Oxaliplatin (D-FOX) in patients with untreated, locally unresectable or metastatic adenocarcinoma of the stomach or gastroesophageal junction (GEJ).

Secondary:

1. To determine the qualitative and quantitative toxicity and reversibility of toxicity of this combination.

Phase II Objectives

Primary:

1. To assess time to cancer progression to D-FOX treatment regimen.

Secondary:

1. To assess response rate to D-FOX treatment regimen.
2. To determine the qualitative and quantitative toxicity and reversibility of toxicity of this combination treatment regimen.
3. Determine overall survival.
4. Perform an exploratory investigation into the effect of D-FOX on phenotypic abnormalities in blood.

DETAILED DESCRIPTION:
Oxaliplatin and 5-FU are chemotherapy drugs that are commonly used to treat certain kinds of cancers. Oxaliplatin interferes with the DNA. 5-FU interferes with cell metabolism. Docetaxel interferes with cell division.

Before you can start treatment on this study, you will have what are called "screening tests". These tests will help the doctor decide if you are eligible to take part in the study. You will be asked questions about your medical history and have a complete physical exam. You will have around 1 tablespoon of blood drawn for routine tests. You will have your height and weight measured. You will have a chest x-ray and an electrocardiogram (ECG - a test that measures the electrical activity of the heart). You will also have a chest x-ray and a computed tomography (CT) scan to check the size and location of the tumor. Women who are able to have children must have a negative blood pregnancy test.

If you are found to be eligible to take part in this study, you will receive treatment with 5-FU as an infusion into a vein using a continuous 24- hour portable pump. This will start on Day 1 and will continue for 48 hours. You will need to carry this pump with you at all times for 48 hours. The pump is about the size of a Sony Walkman®. You will also receive oxaliplatin as an infusion into a vein over 2 hours on Day 1. Docetaxel will be given as an infusion over 60 minutes on Day 1. You will have 12 days to rest between chemotherapy treatments. These drugs may be given to you as an outpatient. Treatment will be repeated on Day 15. Two 14-day treatment periods are called one cycle.

You will be asked to fill out side effect sheets throughout your participation in this research study. You will be asked questions regarding nausea, hair loss, fatigue, meals, and other questions regarding your daily activities. Before each dose of chemotherapy (every 14 days), you will have 1 teaspoon of blood drawn for routine tests.

If the cancer gets worse or you experience intolerable side effects, you will be taken off the study and your doctor will discuss other treatment options with you.

You will be asked to come for a follow-up visit at M.D. Anderson about 2-3 months after treatment ends if possible. At this visit, you will have a full physical, about one tablespoon of blood drawn for routine tests, a chest x-ray, and CT or magnetic resonance imaging (MRI) scans.

This is an investigational study. Oxaliplatin is approved for treatment of colon and rectal cancer but not approved in the US for use in the treatment of gastric cancer. Docetaxel and 5-FU are commonly used drugs for gastric cancer and are commercially available. The combination of these 3 drugs (docetaxel + oxaliplatin + 5-FU) is investigational. A total of up to 106 patients will take part in this study. All will be enrolled at M.D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically documented adenocarcinoma of the stomach or Gastroesophageal Junction (GEJ).
2. Age >18 years;
3. Eastern Cooperative Oncology Group (ECOG) Performance Status 0-1;
4. Chemotherapy: No prior chemotherapy is permitted for metastatic disease. Use of prior chemotherapy in the adjuvant and/or neo-adjuvant setting or as part of a radiosensitization is permitted, provided that the minimum time from completion of such treatment to study entry is at least 12 months;
5. Radiation: Patients may have had prior radiation therapy that has not exceeded 25% of bone marrow reserve provided that they have recovered from the acute, toxic effects of radiotherapy prior to registration. A minimum of 14 days must have elapsed since the end of radiotherapy.
6. Previous Surgery: Previous surgery is permitted provided that wound healing has occurred prior to registration. Minimum of 14 days must have elapsed between a major surgery and start of chemotherapy.
7. At least one target lesion >20 mm (or >10 mm on spiral CT-scan). If indicator lesions are in a previously irradiated field, only a clear disease progression of the irradiated lesion or a new lesion in the previously irradiated field will be accepted
8. Adequate baseline bone marrow, hepatic and renal function, defined as follows: Neutrophils >1.5 * 10*9/L and platelets >100 * 10*9/L; Bilirubin <1.5 * upper limit of the normal range (ULN); aspartate aminotransferase (AST or SGOT) and/or alanine aminotransferase (ALT or SGPT) <2.5 * ULN; Serum creatinine <1.5 * ULN;
9. Patients must give written informed consent to participate in the study.
10. Patients - both males and females - with reproductive potential (ie, menopausal for less than 1 year and not surgically sterilized) must practice effective contraceptive measures throughout the study. Women of child-bearing potential must have a negative pregnancy test (serum or urine) within 14 days prior to registration.

Exclusion Criteria:

1. Concurrent anticancer therapy
2. Pregnant or lactating women
3. History of other prior malignancy except for adequately treated basal cell or squamous cell skin cancer; in situ cervical cancer or malignancy from which the patient has been disease-free for 5 years;
4. Brain metastases
5. Patients with active or uncontrolled infections or with serious illnesses or medical conditions, including patients with a history of chronic alcohol abuse, hepatitis, HIV and/or cirrhosis
6. History of any psychiatric condition that might impair the patient's ability to understand or to comply with the requirements of the study or to provide informed consent.
7. Known hypersensitivity to any of the drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2004-08; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jaffer Ajani, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Result] Blum Murphy MA, Qiao W, Mewada N, Wadhwa R, Elimova E, Takashi T, Ho L, Phan A, Baker J, Ajani J. A Phase I/II Study of Docetaxel, Oxaliplatin, and Fluorouracil (D-FOX) Chemotherapy in Patients With Untreated Locally Unresectable or Metastatic Adenocarcinoma of the Stomach and Gastroesophageal Junction. Am J Clin Oncol. 2018 Apr;41(4):321-325. doi: 10.1097/COC.0000000000000271. PMID 26908161
- See also: UT MD Anderson Cancer Center official website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: September 8, 2004 to August 5, 2009. All recruitment was done at The University of Texas (UT) MD Anderson Cancer Center.
Groups:
- Phase I: Dose Escalation: Phase I: Starting dose of 20mg/m^2 IV Docetaxel over 60 minutes. Dose escalation of Docetaxel in 2.5 mg/m^2 increments until the maximum tolerated dose is determined. 5-Fluorouracil by continuous infusion pump at a dose of 2.2 g/m^2 over 48 hours on Day 1. Oxaliplatin 85 mg/m^2 IV over 120 minutes on Day 1. Treatment was repeated every 14 days (one cycle = 28 days or two 14-day treatments).
- Phase II: Docetaxel MTD 50 mg/m^2: Phase II: Docetaxel 50 mg/m^2 IV over 60 minutes. 5-Fluorouracil by continuous infusion pump at a dose of 2.2 g/m^2 over 48 hours on Day 1. Oxaliplatin 85 mg/m^2 IV over 120 minutes on Day 1. Treatment was repeated every 14 days (one cycle = 28 days or two 14-day treatments).
Period: Overall Study
Arm/Group | Phase I: Dose Escalation | Phase II: Docetaxel MTD 50 mg/m^2
Started | 53 | 45
Completed | 51 | 4
Not Completed | 2 | 41
Not completed — Adverse Event | 2 | 9
Not completed — Disease Progression | 0 | 19
Not completed — Maximal Response | 0 | 6
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Poor Tolerance | 0 | 5

BASELINE CHARACTERISTICS:
Groups:
- Phase I: Phase I: Starting dose of 20mg/m^2 IV Docetaxel over 60 minutes. Dose escalation of Docetaxel in 2.5 mg/m^2 increments until the maximum tolerated dose is determined. 5-Fluorouracil by continuous infusion pump at a dose of 2.2 g/m^2 over 48 hours on Day 1. Oxaliplatin 85 mg/m^2 IV over 120 minutes on Day 1. Treatment was repeated every 14 days (one cycle = 28 days or two 14-day treatments).
- Phase II: Phase II: Docetaxel 50 mg/m^2 IV over 60 minutes. 5-Fluorouracil by continuous infusion pump at a dose of 2.2 g/m^2 over 48 hours on Day 1. Oxaliplatin 85 mg/m^2 IV over 120 minutes on Day 1. Treatment was repeated every 14 days (one cycle = 28 days or two 14-day treatments).
- Total: Total of all reporting groups
Arm/Group | Phase I | Phase II | Total
Number analyzed (Participants) | 53 | 45 | 98
Age, Continuous [Median (Full Range); unit: years] | 55 [24 to 76] | 59 [34 to 79] | 57 [24 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 14 | 26
  Male | 41 | 31 | 72
Region of Enrollment [Number; unit: participants]
  United States | 53 | 45 | 98

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD)
Description: MTD is the highest dose at which 1 or fewer dose limiting toxicities (DLT's) are observed in 6 patients. DLT defined as any non-hematologic grade III/IV or neutropenia-associated (infection or fever treated in the hospital) toxicity attributable to this therapy. Response evaluated after two 14-day treatments of Docetaxel, 5-Fluorouracil and Oxaliplatin (One cycle = 28 days).
Time Frame: 28 days
Measure: Number; unit: mg/m^2
Arm/Group | Phase I
Number analyzed (Participants) | 53
mg/m^2 | 50

2. Primary Outcome: Progression Free Survival
Description: Progression Free Survival (PFS) defined as the time from the first study drug administration until the first day of radiological and/or symptomatic disease progression is documented, or the start of further anticancer therapy or death from any cause, whichever occurs first. Kaplan-Meier curve was used to estimate PFS. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesion.
Time Frame: Assessed from baseline to 30 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase II
Number analyzed (Participants) | 45
months | 6.5 [5.5 to 9.5]

3. Secondary Outcome: Median Overall Survival
Description: Overall survival was defined as the time from the start of treatment until death or last follow-up. Kaplan-Meier curve was used to estimate overall survival.
Time Frame: Up to 30 months
Measure: Median (Full Range); unit: months
Arm/Group | Phase II
Number analyzed (Participants) | 45
months | 11.1 [9.4 to 18.8]

ADVERSE EVENTS:
Time Frame: Adverse event (AE) reporting from time of first intervention, before each dose of chemotherapy (every 14 days) to follow-up 90 days after end of treatment.
Description: NCI Common Terminology Criteria for Adverse Events (CTCAE) version 3.0 utilized for AE reporting.
Arm/Group | Phase I | Phase II
Serious Adverse Events (participants affected / at risk) | 33/53 | 13/45
Other Adverse Events (participants affected / at risk) | 53/53 | 9/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Phase I (N=53) | Phase II (N=45)
Leukopenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Granulocytopenia (Blood and lymphatic system disorders) | 7 (7) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 4 (4) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 11 (11) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (3) | 3 (3)
Vomiting (Gastrointestinal disorders) | 1 (1) | 3 (3)
Anorexia (Gastrointestinal disorders) | 4 (4) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 7 (7) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Hematemesis (Gastrointestinal disorders) | 0 (0) | 1 (2)
Progressive Disease-Brain Mets (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Increasing Abdominal Girth (General disorders) | 0 (0) | 1 (1)
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Increased Bilirubin (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Fever (General disorders) | 0 (0) | 1 (1)
Malaise (General disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Pulmonary Embolism (Vascular disorders) | 0 (0) | 1 (1)
Ventricular Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Gastric Outlet Obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Death (General disorders) | 0/0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I (N=53) | Phase II (N=45)
Leukopenia (Blood and lymphatic system disorders) | 23 (23) | 0 (0)
Granulocytopenia (Blood and lymphatic system disorders) | 15 (15) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 41 (41) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 5 (5) | 0 (0)
Increased ALT (Metabolism and nutrition disorders) | 15 (15) | 0 (0)
Increased AST (Metabolism and nutrition disorders) | 17 (17) | 0 (0)
Increased Creatinine (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 39 (39) | 0 (0)
Dizziness (General disorders) | 13 (13) | 0 (0)
Headache (General disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 43 (43) | 0 (0)
Vomiting (Gastrointestinal disorders) | 27 (27) | 0 (0)
Anorexia (Gastrointestinal disorders) | 37 (37) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 25 (25) | 0 (0)
Taste alteration (Gastrointestinal disorders) | 10 (10) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 18 (18) | 0 (0)
Neuropathy (Nervous system disorders) | 32 (32) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 19 (19) | 0 (0)
Extremity pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0)
Hearing loss (Ear and labyrinth disorders) | 3 (3) | 0 (0)
Tinitis (Ear and labyrinth disorders) | 5 (5) | 0 (0)
Watery eyes (Eye disorders) | 12 (12) | 0 (0)
Blurred vision (Eye disorders) | 2 (2) | 0 (0)
H-F Syndrome (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 26 (26) | 0 (0)
Skin rash (Skin and subcutaneous tissue disorders) | 12 (12) | 0 (0)
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 0 (0)
Neutropenic Fever (General disorders) | 1 (1) | 0 (0)
Vaginal Bleeding (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pedal Edema (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Cytopenias (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Pericardial Effusion (Cardiac disorders) | 0 (0) | 1 (1)
Gastrointestinal Bleeding (Gastrointestinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes